CLINICAL TRIAL: NCT00944840
Title: A Trial of Intermittent Preventive Treatment and Home Based Management of Malaria in a Rural Area of The Gambia
Brief Title: Intermittent Preventive Treatment (IPTc) and Home Based Management of Malaria (HMM)in The Gambia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCC 1124
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Intermittent Preventive Treatment; Home based management of malaria
MeSH Terms: conditions — Malaria | interventions — Amodiaquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SP and amodiaquine (Active Comparator): Study subjects received intermittent preventive treatment with SP plus amodiaquine.
  Interventions: Drug: SP plus amodiaquine
- SP placebo plus amodiaquine placebo (Placebo Comparator): Intermittent preventive treatment with SP placebo and amodiaquine placebo
  Interventions: Drug: SP placebo plus amodiaquine placebo

INTERVENTIONS:
Drug: SP plus amodiaquine — SP plus amodiaquine or placebo at monthly interval during September, October and November
  Other Names: Camoquin; Fansidar
  Arms: SP and amodiaquine
Drug: SP placebo plus amodiaquine placebo — monthly treatment with amodiaquine and SP or placebo during September, October and November
  Arms: SP placebo plus amodiaquine placebo

SUMMARY:
Malaria in African countries remains an important cause of mortality and morbidity among young children. The global malaria control strategies include prompt treatment with an effective antimalarial drug, vector control using ITNs or curtains, indoor residual spraying (IRS), and intermittent preventive treatment. However, individually these interventions provide only imperfect protection. Thus, there is a need to investigate whether additional control measures provide added benefit in reducing mortality and morbidity. Therefore, 1312 children under 5 years of age living in villages and hamlets near Farafenni, The Gambia, which form part of the rural Farafenni Demographic Surveillance system (FDSS) in North Bank Region(NBR) were randomly allocated to receive IPTc or placebo from village health workers based in primary health care villages. Treatment with a single dose of sulfadoxine /pyrimethamine plus three doses of amodiaquine or placebo was given to all study subjects at monthly intervals on three occasions during the months of September, October and November. In addition, VHWs were trained to administer treatment with coartem to children if they develop symptoms compatible with malaria during the malaria transmission season. The primary end point was the incidence of clinical attacks of malaria detected during the study.

DETAILED DESCRIPTION:
Goals and Objectives

1. The goal of this project was to determine the degree to which morbidity from malaria can be prevented in children who receive intermittent preventive treatment(IPTc) with SP plus amodiaquine and home based management of malaria with Coartem by village health worker during 2008 malaria transmission season.
2. The objective of the project was to conduct an individually randomized trial of IPTc in children who receive HMM in North Bank Region an area where malaria transmission is highly seasonal. This trial will determine whether IPTc adds significant benefit to HMM.

   The study was undertaken in a group of 42 villages and hamlets near Farafenni. The villages ranged in size from 46 to 1250 inhabitants. The total population of the rural FDSS catchment area was about 17 000 and that of children under 5 years of age was about 3000. The area has one general hospital, three health centres and two private healthcare clinics. There are 18 rural primary health care (PHC) villages in the study area. PHC villages, each with a population over 400, have mainly been selected plus, occasionally, others located in relatively isolated areas. In all villages, village health workers (VHWs) and traditional birth attendants (TBAs) are selected by the Village Development Committee (VDC) and given 6 to 8 weeks of training with a standardised curriculum on how to treat common conditions such as uncomplicated malaria, ARI, diarrhoeal diseases and minor injuries. Thus, VHWs function as primary health care providers for minor illnesses and injuries for all ages. In addition, the VHW are expected to work as a community-based health educator. TBAs functioned as birth attendants, family planning distributors and health educators. Both TBAs and VHWs were expected to refer serious cases to the local health facility for management. VHWs and TBAs are supervised by Community Health Nurses who oversee circuits of 4 to 10 PHC villages. All rural settlements also have a Medical Research Council(MRC) Village Reporter who carries out sensitization for MRC activities. The bednet coverage in NBR was estimated to be 50%. However, during the study, details of bed net usage by the community were assessed.

   Recruitment and randomization:

   The study was carried in collaboration with the EPI unit of the Department of State for Health, National Malaria Control Programme and NBR District Health Team. During the preparatory phase of the study, the design and objectives of the study were discussed extensively with the NBR District Team and all health care providers working in the study area. The study team visited all the villages in the study area to explain the objectives of the trial to village elders, opinion leaders, and heads of women's groups, village health workers and traditional birth attendants. This was followed by village meetings, at which the entire community was invited to participate. During these meetings, agreement to participate in the study was obtained from the villagers. In addition, parents or guardians of prospective study subjects in the right age group were visited at home and they were provided with flyers in English and the appropriate local language (Mandinka, Wollof or Fula). Written informed consent was obtained from the parent(s) or guardian(s) before a child was enrolled in the study. Enrolled subjects were provided with a treatment card stamped with a label carrying their name and study number to facilitate identification at each contact.

   Individual randomization was carried out. Study subjects were allocated to receive IPTc plus HMM or HMM alone.

   IPTc and malaria treatment:

   Study children received their monthly treatment from a VHW based in a PHC village. The VWH distributed the trial medication at a central point (usually a health post) during the first 10 days of the month during September, October and November. Mothers and carers were asked to bring their children to the central point during the morning when the VWH was available to distribute the drugs. When a child presented to the central point for medication, the VHW identified the study subject using the treatment card held by the mother and matched the information on the treatment card with that on his register. When he was satisfied that he had correctly identify the study subject, the correct dosage of the trial medication was given to the study subject. In non-PHC villages, mothers were asked to bring their children to their nearest PHC village to receive IPT during the transmission season.

   The first dose of treatment was taken under direct supervision of the VHW and the remaining two doses were given to the mother or guardian of the child with clear instructions on how to administer the drugs.

   At the end of the malaria transmission season, the total number of complete treatment doses each child in the trial had taken was recorded. Compliance was checked on a rolling basis throughout the study by assessing the number of correct doses of medication received.

   Malaria treatment and morbidity surveillance during the rainy season Passive surveillance for malaria was maintained throughout the transmission season. VHW were instructed to treat febrile illnesses suggestive of malaria with coartem . Parents/guardians were encouraged to take their child to the VHW at any time the child became unwell. One field worker was attached to 2-3 village health workers during the surveillance period. The role of the field worker was to prepare a thick blood film from children scheduled for treatment by the VHW with coartem for subsequent confirmation of the diagnosis. VHWs were asked to keep records of children treated for malaria. In addition, they were asked to refer children who failed to improve on treatment and those with danger signs to the nearest health centre or AFPRC Hospital for further evaluation and management.

   Any death of a study child was investigated within a month of death using the post-mortem questionnaire technique.

   Cross-sectional survey:

   In December, at the end of the malaria transmission season, a cross-sectional survey of all the children enrolled in the study was undertaken in all the villages. Information was obtained on demographics, bed net usage, a clinical history was obtained and a physical examination performed, including abdominal palpation for splenomegaly and measurement of height, weight and axillary body temperature. A finger-prick blood sample was obtained from all the children taking part in the cross-sectional survey for preparation of blood films, a filter paper sample and determination of the haemoglobin level.

   Definitions

   The following definitions were used during the course of the study.

   Clinical malaria. The primary definition of malaria required:
   1. the presence of fever (axillary temperature > 37.5 C) or a history of fever in the past 24 hours,
   2. the absence of any other obvious cause of the fever,
   3. the presence of P. falciparum asexual parasitemia above a threshold value of 5,000 parasites per ul (a threshold shown previously to be of value in differentiating symptomatic malaria from other illnesses associated with co-incidental parasitemia).

   A secondary definition of malaria required only the presence of P. falciparum parasitemia at any density.

   Severe malaria. Severe malaria was defined according to the WHO criteria

   Anemia. Anemia was defined as a haemoglobin(Hb) concentration <11 g/dl, moderate anemia as a Hb concentration < 8 g/dL and severe anemia as an Hb concentration < 5 g/dl.

   End-points:

   Primary endpoint :

   Malaria incidence (the number of study subjects seen at the OPD clinic with clinical malaria that meet the primary case definitions as indicated above during the surveillance period).

   Secondary endpoints :
   1. Malaria incidence (the number of study subjects seen by the VHW with clinical malaria that meet the secondary case definitions as indicated above during the surveillance period).
   2. the incidence of severe malaria as defined above,
   3. the incidence of anaemia among children seen at a hospital or health centre,
   4. the prevalence of parasitaemia at the end of malaria transmission season cross-sectional survey,
   5. the prevalence of anaemia at the end of malaria transmission season cross-sectional survey,

   (d) the incidence of all cause hospital admissions,

   (e) the incidence of hospital admissions due to malaria,

   (f) Coverage with IPTc as measured by the following indicators:
   * the proportion of children who received three IPT courses on schedule;
   * the proportion of children who received partial or off-schedule IPT courses
   * the proportion of children with no IPT.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 3 months and 59 months at enrolment.
2. Informed consent obtained from parents or legal guardians.
3. No current participation in another malaria intervention trial
4. Permanent residence in the study area with no intention of leaving during the surveillance period.

Exclusion Criteria:

1. Previous adverse reaction to treatment with SP, amodiaquine or Coartem. If this is unknown, then a history of allergic reaction to any drug.
2. Temporary residence in the study area
3. Lack of informed consent
4. Presence of a severe, chronic illness such as severe malnutrition or AIDS, likely to interfere with evaluation of the trial results.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1312 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Malaria incidence (the number of study subjects seen at the OPD clinic with clinical malaria during the surveillance period). | During the surveillance period (September to December 2008)

SECONDARY OUTCOMES:
prevalence of parasitaemia at the end of malaria transmission season in December 2008 | December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Kalifa Bojang, MD, PhD, Principal Investigator — MRC Laboratories
Locations (1):
- Farafenni Field Station, MRC Laboratories, Farafenni, North Bank Division, The Gambia

REFERENCES:
- [Derived] Sesay S, Milligan P, Touray E, Sowe M, Webb EL, Greenwood BM, Bojang KA. A trial of intermittent preventive treatment and home-based management of malaria in a rural area of The Gambia. Malar J. 2011 Jan 7;10:2. doi: 10.1186/1475-2875-10-2. PMID 21214940